CLINICAL TRIAL: NCT06196372
Title: The Effect of Online Cognitive Awareness-Based Nursing Support for Premenopausal Women on Vasomotor Symptoms, Stress and Quality of Life
Brief Title: Online Cognitive Awareness-Based Nursing Support for Premenopausal
Acronym: (MenoMind)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Fatma Aslan Demirtaş, Research Assistant, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BandırmaOnyediEylulU-FAD-01
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Pre-Menopause; Irregular Menstruation
Keywords: Pre-menopause,; Mindfulness; Vasomotor; Stress; Quality of life
MeSH Terms: conditions — Menstruation Disturbances

STUDY DESIGN:
Intervention Model Description: The design of this study is a randomized controlled experimental study with a single-blind pretest-posttest control grou
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention (Experimental): An online mindfulness nursing support program (MenoMind) was applied to this group for 8 weeks and lasting an average of 50 minutes.
  Interventions: Other: MenoMind intervention group
- Control (No Intervention): The control group received no intervention and the women were left to routine clinical care.

INTERVENTIONS:
Other: MenoMind intervention group — To implement the MenoMind program, the women in the initiative group were divided into groups of 4-5 according to their convenient days and hours, and it was done via the Zoom© program. MenoMind program was carried out via video on WhatsApp© program for women who could not or did not want to use the Zoom© program. The researcher provided support to the women for eight weeks, in different groups, 2-3 days a week and at different times, depending on their availability. Each session is approximately 50 minutes. lasted. In addition, make-up sessions were organized for women who could not attend the sessions for various reasons or had difficulty complying with the program (day/date).
  Arms: Experimental: Intervention

SUMMARY:
This randomized controlled study was conducted at Istanbul University-Cerrahpaşa Cerrahpaşa Medical Faculty Hospital between 16.05.2022-30.06.2023. Research data were collected at the gynecology outpatient clinic. The sample of the study consisted of 74 (37-intervention, 37-control) premenopausal women who met the inclusion criteria and were placed by randomization. The data of the study were collected using "Personal Information Form, Mindful Attention Awareness Scale (MAAS), Visual Analogue Scale for Vasomotor Symptoms (VAS), Perceived Stress Scale (PSS) and Menopause-Specific Quality of Life Scale (MENQOL)". First, the pretests of the study were applied to women in the intervention and control groups. Afterwards, women in the intervention group underwent the MenoMind program for eight weeks, and women in the control group were left with routine clinical care. In the eighth week of the research, the "MenoMind Evaluation Form" was applied to the women in the intervention group to evaluate the MenoMind program. One month after the study was completed, post-tests were performed on the intervention and control groups.

DETAILED DESCRIPTION:
METHOD Purpose of the research This study aims to examine the effect of online cognitive awareness-based nursing support (MenoMind) for premenopausal women on vasomotor symptoms, stress and quality of life.

Type of research This study was planned as a randomized controlled experimental study. The study was conducted according to CONSORT guidelines.

Hypotheses of the research Hypothesis 1: MenoMind program increases the conscious awareness level of premenopausal women.

Hypothesis 2: The MenoMind program reduces vasomotor symptoms of premenopausal women.

Hypothesis 3: The MenoMind program reduces the stress level of premenopausal women.

Hypothesis 4: MenoMind improves the quality of life of premenopausal women.

Population and sample of the research The universe of the research; The sample consisted of premenopausal women with menstrual irregularities who applied to the Gynecology Polyclinic of Istanbul Cerrahpaşa Medical Faculty Hospital for control purposes.

The power of the study was calculated in the G*Power program, taking Perceived Stress Scale as the main parameter for the sample of the study. It was planned to form a sample of 74 premenopausal women, whose number was higher according to the G*Power analysis results.

Implementation of research The researcher attended the training program for the implementation of the Mindflness Stress Reduction Program, received a hereditary certificate and started researching as a practitioner.Afterwards, an online mindfulness -based nursing support program (MenoMind) was created in accordance with the Mindfulness Stress Reduction Progra. The MenoMind program is an eight-week program suitable for online conditions for premenopausal women and lasts an average of 50 minutes a week. "MenoMind" and "Healthy Menopause: Every Woman's Right" training booklets were created by researchers for the MenoMind program. The "MenoMind" training booklet is a guide for women in the initiative group. The "MenoMind" training booklet includes preliminary preparation for the sessions, the purpose of the sessions, information about the applications to be applied in the sessions, evaluation questions and homework to evaluate the session after the sessions throughout the MenoMind program. The "Healthy Menopause: Every Woman's Right" training booklet provides women with information about what they will experience during the menopause period. It was prepared to inform them about the symptoms and how to cope with these symptoms. The training booklet "Healthy Menopause: Every Woman's Right" was planned to be sent via WhatsApp© to women in the intervention group during the week of the 1st Session, and to women in the control group after the final test was performed. These training booklets were planned to be sent to the women in the intervention group via WhatsApp©. Before starting, it was sent to faculty members who are experts in their fields to get their opinions and suggestions. The final version of the training booklets was created in line with the suggestions made by the faculty members.

Preliminary tests of the research were first applied to women in the intervention and control groups who accepted the research and met the inclusion criteria (being able to read and write, being able to use the internet, having a device that can use the internet, not having a diagnosed psychiatric disease, not having a chronic disease, not using hormone replacement therapy, age 40 and above and having symptoms of menstrual irregularity, having vasomotor symptoms). Afterwards, the researcher divided the women in the intervention group into groups of 4-5 according to the appropriate days and hours to implement the MenoMind program, and it was done via the Zoom© program. MenoMind program was carried out via video on WhatsApp© program for women who could not or did not want to use the Zoom© program. The researcher provided support to the women for eight weeks, in different groups, 2-3 days a week and at different times, depending on their availability. Each session is approximately 50 minutes lasted. In addition, make-up sessions were organized for women who could not attend the sessions for various reasons or had difficulty complying with the day/date schedule. After the MenoMind program application started, a WhatsApp message was sent to women on the days of the sessions to remind them of the session time and the necessary preparations for the session. After each session of the eight-week program, women were asked to repeat the MenoMind applications and were given weekly homework for them. Session recordings were sent to women and they were given a "MenoMind" training booklet to help them with weekly homework. When the program started each week, the first thing that was discussed was homework. At the end of the session in the eighth week of the MenoMind program, each woman was interviewed and the "MenoMind Evaluation Form" was applied to evaluate the program content and the researcher's application technique. One month (4 weeks) after completing the application, the tests were administered to the women in the intervention group for the last time.

During the implementation of the study, no intervention was applied to the control group and the women were left to routine clinical care. At the end of the research, in accordance with the principle of equality, the women in the control group were given a "Healthy Menopause: Every Woman's Right" educational booklet.

Data Evaluation Data were analyzed using SPSS (Statistical Package for the Social Sciences) 23.0 (IBM Corp., Armonk, NY, USA). Mean, standard deviation, frequency, number and percentage were used to determine the descriptive characteristics of the participants. Shapiro-Wilk test was used to evaluate normal distribution. Dependent groups t test was used for intragroup comparisons, and independent sample t test was used for intergroup comparisons. Relationships between continuous variables were examined with Pearson correlation analysis. The results were evaluated within the 95% confidence interval, with significance below p<0.05.

Ethical Aspects of the Study The study was conducted in accordance with the principles of the Declaration of Helsinki. Ethical permission for the research was obtained from Istanbul University Cerrahpaşa Non-Interventional Clinical Research Ethics Committee (Date and number: 13.05.2022 -2022/35), Institutional permission for the research was obtained from Istanbul University- Cerrahpaşa, Cerrahpaşa Faculty of Medicine, Department of Gynecology and Obstetrics. Taken from. Women were informed about the research and their consent was obtained in accordance with the "Informed Volunteer Consent Form".

ELIGIBILITY:
Inclusion Criteria:

* Being able to read and write,
* Being able to use the internet,
* Having a device that can use the internet (such as a smartphone or computer),
* Not having a diagnosed psychiatric disease,
* Not having a chronic disease
* Not using hormone replacement therapy,
* Age 40 and above and having symptoms of menstrual irregularity,
* Receiving an average score of two or more from Menopause-Specific Quality of Life Scale,
* Scoring three or more on the Visual Analogue Scale for Vasomotor Symptoms

Exclusion Criteria:

* There are situations that prevent the exercises from being performed,
* Participating in a mindfulness training program before.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The groups were created by women in the premenopausal period.
Enrollment: 74 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | 5th minute
  The personal information form, created in line with the literature, aims to determine the socio-demographic characteristics of women in the premenopausal period; It is a form consisting of 13 items containing descriptive information specific to the individual (age, education, marital status, employment status, income level, vasomotor symptoms, smoking status and regular exercise status).

SECONDARY OUTCOMES:
Mindful Attention Awareness Scale (MAAS) | 5th minute
  MAAS was developed by Brown and Ryan in 2003. The scale is a six-point Likert type (1 - almost always, 4 - almost never) and consists of 15 items. A single total score is obtained in MAAS. The lowest score that can be obtained from the scale is 15 and the highest score is 90.
Visual Analog Scale for Vasomotor Symptoms (VAS) | 2th minute
  VAS allows numerical measurement of values that cannot be measured numerically. These parameters are written at both ends of a 100 mm line to determine the severity of hot flashes, sweating and night sweats. The woman is asked to indicate the suitability of her situation by pointing, drawing a line, or placing a dot on this line. By choosing the appropriate value for women, the severity of hot flashes, night sweats and sweating are determined. Evaluation of VAS is made by taking the average of the scores obtained.
Perceived Stress Scale (PSS) | 5th minute
  PSS, Cohen et al. It was developed by in 1983. The five-point Likert type scale (0 - never, 4 - very often) consists of 14 items. The scale has two subscales. Perception of stress/discomfort (questions 1, 2, 3, 7, 11, 12, 14) and perception of insufficient self-efficacy (questions 4, 5, 6, 8, 9, 10, 13). The scale has no cut-off point. It is understood that as the score of the scale increases, the person's perception of stress increases.
Menopause-Specific Quality of Life Scale (MENQOL) | 10th minute
  MENQOL, Hilditch et al. It was developed by in 1996. The Likert type scale consists of 29 items. The scale total is calculated using the average score. The preliminary lowest score that can be obtained from the scale is 0, and the highest score is 6. A score of "0" indicates that there is no problem regarding the issue, a score of "1" indicates that the problem exists but is not disturbing, and scores between "2-6" indicate the severity and increasing degrees of the existing problem. The scale consists of four areas. They are the vasomotor domain (questions 1-3), the psychosocial domain (questions 4-10), the physical domain (questions 11-26) and the sexual domain (questions 27-29).

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Aslan Demirtaş, Msc, Principal Investigator — Bandırma Onyedi Eylül University
Locations (1):
- Istanbul University-Cerrahpaşa Cerrahpaşa Medical Faculty Hospital between, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No